CLINICAL TRIAL: NCT02669394
Title: Reshaping the Path of Vascular Cognitive Impairment With Resistance Training
Brief Title: Reshaping the Path of Vascular Cognitive Impairment (VCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-00972
Record Dates: First submitted 2016-01-14; First posted 2016-02-01 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Transient Ischemic Attack; Vascular Cognitive Impairment; Subcortical Vascular Dementia
MeSH Terms: conditions — Ischemic Attack, Transient; Dementia, Vascular | interventions — Resistance Training; Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistance Training (RT) (Experimental): The RT program will be a twice-weekly program. A pressurized air system and free weights will be used . The pressurized air system exercises will consist of biceps curls, triceps extension, seated row, latissmus dorsi pull downs, leg press, hamstring curls, and calf raises. Other exercises, with free weights, will include mini-squats, mini-lunges, and lunge walks. The intensity of the training stimulus will initially be at 50% to 60% of 1 repetition maximum (RM) as determined at week two, and progress to 75% to 85% of 1-RM at a work level of 6 to 8 repetitions (2 sets) by week four. The training stimulus will be increased using the 7 RM method.
  To meet the public health mandates of COVID-19, when it is necessary, training will occur at home, with the use of a set of resistance bands of various weights. Participants will be provided access to instructional videos either by YouTube or DVD. They will be called on a weekly basis to monitor progress and compliance.
  Interventions: Behavioral: Resistance exercise training
- Stretching and Relaxation (CON) (Active Comparator): The CON program will be a twice-weekly program. The CON group will consist of stretching exercises, basic core-strength/kegal exercises, and relaxation techniques. Other than bodyweight, no additional loading (e.g., hand weights, resistance bands, etc.) will be applied to any of the exercises.
  To meet the public health mandates of COVID-19, when it is necessary, training will occur at home. Participants will be provided access to instructional videos either by YouTube or DVD. They will be called on a weekly basis to monitor progress and compliance.
  Interventions: Behavioral: Control: stretching and relaxation program

INTERVENTIONS:
Behavioral: Resistance exercise training — Twelve months of twice-weekly resistance training program that will gradually progress in intensity. Each training session will be 60 minutes (10 minutes of warm-up, 40 minutes of training, and 10 minutes of cool-down).
  Other Names: RT Program
  Arms: Resistance Training (RT)
Behavioral: Control: stretching and relaxation program — Twelve months of twice-weekly stretching and relaxation program that includes stretches, deep breathing and relaxation techniques, general core control exercises, and general posture and health education. Each session will be 60 minutes.
  Other Names: CON Program
  Arms: Stretching and Relaxation (CON)

SUMMARY:
The investigators will conduct a proof-of-concept randomized controlled trial study to provide preliminary evidence of efficacy of a resistance exercise training program for maintaining white matter health and improving cognitive function in older adults with vascular cognitive impairment, defined as the presence of cognitive impairment combined with cerebral small vessel disease, compared with a stretch and relaxation program.

DETAILED DESCRIPTION:
A total of 88 adults with vascular cognitive impairment will be randomized to either a 12-month twice-weekly resistance training program or stretch and relaxation program. There will be three measurement sessions: baseline, 6 months (midpoint of intervention period), and 12 months (end of intervention period).

ELIGIBILITY:
Inclusion Criteria:

The study will specifically recruit individuals who fulfill the diagnostic criteria for SIVCI -- the presence of both cognitive impairment and small vessel ischaemic disease.

Specifically, individuals must meet the following inclusion criteria:

1. Montreal Cognitive Assessment (MoCA) score less than 26 at screening;
2. MMSE score of = or > 20 at screening;
3. Community-dwelling;
4. Lives in Metro Vancouver;
5. Able to comply with scheduled visits, treatment plan, and other trial procedures;
6. Must be able to read, write, and speak English in which psychometric tests are provided with acceptable visual and auditory acuity;
7. Stable on a fixed dose of cognitive medications (e.g., donepezil, galantamine, rivastigmine, memantine, etc.) that is not expected to change during the 12-month study period, or, if they are not on any of these medications, they are not expected to start them during the 12-month study period;
8. Provide a personally signed and dated informed consent document indicating that the individual (or a legally acceptable representative) has been informed of all pertinent aspects of the trial. In addition, an assent form will be provided at baseline and again at regular intervals;
9. Able to walk independently; and
10. Must be in sufficient health to participate in study's aerobic-based exercise training program. This will be based on medical history, vital signs, physical examination by study physicians, and written recommendation by family physician indicating individual's appropriateness to participate in an aerobic-based exercise training program.

Exclusion Criteria:

1. Absence of relevant small vessel ischaemic lesions on an existing brain computed tomography (CT) or MRI;
2. Diagnosed with another type of dementia (e.g., AD) or other neurological conditions (e.g., multiple sclerosis, Parkinson's disease, etc.) that affects cognition and mobility;
3. Diagnosed previously with a genetic cause of SIVCI (e.g., CADASIL);
4. At high risk for cardiac complications during exercise and/or unable to self-regulate activity or to understand recommended activity level (i.e., Class C of the American Heart Risk Stratification Criteria);
5. Participating in regular RT in the last six months;
6. Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility;
7. Taking medications that may negatively affect cognitive function, such as anticholinergics, including agents with pronounced anticholinergic properties (e.g., amitriptyline), major tranquilizers (typical and atypical antipsychotics), and anticonvulsants (e.g., gabapentin, valproic acid, etc.); or
8. Individual who plans to participate or is enrolled in a clinical drug trial concurrent to this study.
9. Unable to meet the specific scanning requirements of the UBC 3T MRI Research Centre. Specifically, we will exclude anyone with: pacemaker, brain aneurysm clip, cochlear implant, recent surgery or tattoos within the past 6 weeks, electrical stimulator for nerves or bones, implanted infusion pump, history of any eye injury involving metal fragments, artificial heart valve, orthopedic hardware, other metallic prostheses, coil, catheter or filter in any blood vessel, ear or eye implant, bullets, or other metallic fragments.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function as measured by Alzheimer's Disease Assessment Scale Cognitive Subscale Plus (ADAS-Plus) | Baseline, 6 months, and 12 months
  ADAS-Cog 13 Plus additional cognitive tests
Change in white matter health as measured by total white matter lesion volume | Baseline to 12 months
  White matter hyperintensity volume in mm3

SECONDARY OUTCOMES:
Executive functions as measured by standard neuropsychological tests | Baseline, 6 months, and 12 months
Arterial stiffness as measured by carotid-femoral arterial pulse-wave velocity (PWV) (subset only) | Baseline and 12 months
Cardiometabolic risk factors as measured by blood panel (subset only) | Baseline, 6 months, and 12 months
Cardiometabolic risk factors as measured by body mass index | baseline, 6 months, and 12 months
Cardiometabolic risk factors as measured by waist to hip ratio | baseline, 6 months, and 12 months
Physiological falls risk as measured by the Physiological Profile Assessment | baseline, 6 months, and 12 months
Mobility and balance as measured by the Short Physical Performance Battery | baseline, 6 months, and 12 months
Mood as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) | baseline, 6 months, and 12 months
Quality of life as measured by the Medical Outcomes Study Short Form-6D (SF-6D) | baseline, 6 months, and 12 months
White matter integrity as measured by diffusion tensor imaging | baseline and 12 months
Myelin plasticity as measured by multicomponent relaxation imaging | baseline and 12 months
Memory as measured by standard neuropsychological tests | baseline, 6 months, and 12 months
Upper body strength as measured by grip strength | baseline, 6 months, and 12 months
Lower body strength as measured by 30 sec sit to stand test | baseline, 6 months, and 12 months
Functional capacity as measured by 6 minute walk test | Baseline, 6 months, 12 months
Neurotrophic factors in blood: IGF-1, BDNF, VEGF (subset only) | Baseline, 6 months, 12 months
Self-reported physical activity as measured by the PASE questionnaire | Monthly
NIH Cognitive Toolbox | Baseline, 6 months, 12 months
Isokinetic strength of the lower limb (subset only) | Baseline, 6 months, 12 months
Functional connectivity using resting state fMRI (subset only) | Baseline and 12 months
Health resource utilization | Baseline and every 3 months
Prospective falls via monthly falls calendars | Monthly
Mobility using Timed up and Go Test | Baseline, 6 months, 12 months
Dual-task ability using dual-task timed up and go test | Baseline, 6 months, 12 months
Dual task gait using Gaitrite mat (subset only) | Baseline, 6 months, 12 months
Cognitive function using ADAS-Cog 13 | Baseline, 6 months, 12 months
Dominant quad isometric strength using a strain gauge | Baseline, 6 months, 12 months
Hypothalamic-pituitary-adrenal axis activity using saliva samples (i.e., cortisol) (subset only) | Baseline, 6 months, 12 months
Regional brain volumes using structural MRI | Baseline and 12 months
Selected Pro- and anti-inflammatory cytokines in blood (subset only) | Baseline, 6 months, and 12 months
  IFN-alpha, IL-1 alpha, IL-4, IL-6, IL-10, IL-12p70, IL-13, IL-17, TNF-alpha, Rantes, CXCL1, IL-18, TGF-B
Telomere Length (subset only) | Baseline, 6 months, and 12 months
Sleep quality as measured by MW8 | Baseline, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, PT, Principal Investigator — University of British Columbia; John Best, PhD, Principal Investigator — University of British Columbia; Jennifer Davis, PhD, Principal Investigator — University of British Columbia; Charlie Goldsmith, PhD, Principal Investigator — Simon Fraser University; Ging-Yuek Robin Hsiung, MD, PhD, Principal Investigator — University of British Columbia; Roger Tam, PhD, Principal Investigator — University of British Columbia; Thalia Field, MD, Principal Investigator — University of British Columbia; Kenneth Madden, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balbim GM, Boa Sorte Silva NC, Falck RS, Kramer AF, Voss MW, Liu-Ambrose T. 24-hour activity cycle behaviors and gray matter volume in mild cognitive impairment. Alzheimers Dement. 2025 Jul;21(7):e70496. doi: 10.1002/alz.70496. PMID 40693459
- [Derived] Liu-Ambrose T, Dao E, Crockett RA, Barha CK, Falck RS, Best JR, Hsiung GR, Field TS, Madden KM, Alkeridy WA, Boa Sorte Silva NC, Davis JC, Ten Brinke LF, Doherty S, Tam RC. Reshaping the path of vascular cognitive impairment with resistance training: a study protocol for a randomized controlled trial. Trials. 2021 Mar 18;22(1):217. doi: 10.1186/s13063-021-05156-1. PMID 33736706